CLINICAL TRIAL: NCT04029870
Title: Psychological déterminants of the Therapeutic Observance of Osteoporotic Patients
Brief Title: Psychological Determinants of the Therapeutic Observance of Osteoporotic Patients
Acronym: OSTEOPSY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-02Obs-CHRMT
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Osteoporosis; adherence to therapy; psychological determinants; self regulation model
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Osteoporosis is a skeletal pathology characterized by decreased bone mass and deterioration of bone tissue. This pathology affects predominantly women, which is estimated that 40% of them will suffer an osteoporotic fracture. The incidence of osteoporosis, thus representing a major public health problem where osteoporotic fractures have a higher incidence than those combined with cardiovascular disease and breast cancer (INSERM, 2016; WHO 2008). It causes traumatic fractures that have the effect of dependence and loss of functional autonomy associated, in terms, with the risk of a reduction in life expectancy. The management of osteoporosis therefore becomes an issue for rheumatologists. The latter involves both compliance with hygienic-Dietetic measures (such as calcium intake, physical activities, prevention of falls...) and medicated treatments whose action is intended, for some, to block bone destruction or, for others to stimulate bone formation. The efficacy of drug treatments is now proven, these treatments are however profitable only if the therapeutic adherence of the patients is maximal. However, rheumatologists and researchers generally find an average rate of 70% enrolment after 6 months of treatment, most often lowered to 50% after 12 months of treatment, thus increasing fractures.

On the other hand, the literature informs the medical and educational aspects of the problem of non-observance in osteoporotic patients, but curiously, it does not say anything of the psychological aspects likely to be linked to these behaviors of non-adherence to therapy.

The objective of this thesis work is to take an interest in the underlying psychological determinants that may explain the behaviour of adherence and/or non-adherence of osteoporotic patients.

ELIGIBILITY:
Inclusion Criteria:

* Be treated with an anti-osteoporotic drug for at least three months
* Mastering the French language orally and in writing
* Have obtained the patient's oral agreement to participate in the research
* Present post-menopausal osteoporosis
* Present a densitometric osteoporosis with a T-score (-2.5) treated medically per OS (example: biphosphonates) or by subcutaneous injection (example: prolia)
* Present a history of severe osteoporotic fractures after falls of its height.

Exclusion Criteria:

* Present a psychiatric history
* Present an intellectual disability
* Present major cognitive disorders related to neurodegenerative disease or other nervous system disorders.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with post-menopausal osteoporosis
Study Population: The study will focus on a sample of 200 post-menopausal osteoporotic patients.
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Adherence to therapy | Day 1
  The influence of psychological emission on the therapeutic adherence is measured with an adherence scale (EGOMAC) which includes 3 items: drugs observance, hygiene compliance and dietary restrictions. The item are scored on a 4-point scale with 1-strongly disagree; 2-disagree, 3-agree and 4-fully agree.

SECONDARY OUTCOMES:
Adherence to therapy | Year 1
  The influence of psychological emission on the therapeutic adherence is measured with an adherence scale (EGOMAC) which includes 3 items: drugs observance, hygiene compliance and dietary restrictions. The item are scored on a 4-point scale with 1-strongly disagree; 2-disagree, 3-agree and 4-fully agree.
Perception of disease | day 1
  with the validated Brief Illness Perception Questionnaire.The Brief IPQ has nine items rated on a scale from 0 (minimum) to 10 (maximum). The first five assess cognitive perceptions such as effect on life; duration of illness control over illness; beliefs about the effectiveness of treatment, and experience of symptoms. Items 6 and 8 assess emotional aspects to include concern about illness and a multifaceted question about mood. Item 7 assesses degree of understanding of the illness. The final item is open-ended asking respondent to rank the 3 most impotant factors causing their illness.
Perception of treatment | day 1
  Wit the Beliefs about Medicines Questionnaire which comprises 18 items which assesses medication beliefs in general and in specific conditions allowing for the investigation of the overall perceptions of medication in general as well as perceptions of medication in their chronic disease. The item are scored on a 5 point Likert scale with scores ranging from 4 to 20.
Anxiety | day 1
  Anxiety is measured with the Hospital Anxiety and Depression Scale composed of 14 items, seven items for the anxiety subscale and seven for the depression subscale. Each item is scored on a response-scale with four alternatives ranging between 0 and 3. For both subscale, score of less than 7 indicates non-cases; between 8 and 10: mild; between 11 and 14: moderate and between 15 and 21: severe.

CONTACTS AND LOCATIONS:
Locations (1):
- CHR Metz Thionville, Metz, Moselle, France